CLINICAL TRIAL: NCT06216964
Title: Time to Clearance of Chlamydia Trachomatis and Neisseria Gonorrhoeae RNA After Treatment: a Prospective Cohort Study
Acronym: DECHLAGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9188
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Chlamydia Trachomatis; Neisseria Gonorrhoeae; Uncomplicated Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chlamydia trachomatis (CT) and/or Neisseria gonorrhoeae (NG) NAAT(s) — Test every week after the start of treatment, until NAAT negativation and up to a maximum of 4 weeks

SUMMARY:
The aim of this study is to evaluate the negativation time of chlamydial and gonococcal PCRs after treatment for urogenital, oropharyngeal and anal infections.

ELIGIBILITY:
Inclusion Criteria:

* - Patients attending the Trait d'Union department at the Nouvel Hôpital Civil for PrEP consultations, AES or HIV infection.
* Over 18 years of age
* Male or female
* Who have had an uncomplicated CT and/or NG infection treated with currently recommended therapies (Ceftriaxone 500mg DU for NG infections, Doxycycline 200mg per day for 1 week for rectal CT infections and Azithromycin 1g DU or Doxycycline 7 days for other CT infections).
* Subject affiliated to a social health insurance scheme
* Subject able to understand the aims and risks of the research and to give dated and signed informed consent

Exclusion Criteria:

* - Complicated CT and/or NG infections: epididymitis, prostatitis, upper genital infection, extra-genital involvement (keratoconjunctivitis, arthritis, skin involvement, Fiessinger-Leroy-reiter syndrome, Fitz-Hugh-Curtis syndrome).
* Interfering treatments and associated diseases: Severe immunosuppression (HIV infection with CD4 less than 200/mm3, chemotherapy in the last 6 months, active haemopathy, congenital immune deficiency, immunosuppressive treatment including corticosteroid therapy for more than 4 weeks or organ transplant.
* Impossibility of giving the subject informed information (subject in an emergency situation, difficulties in understanding the subject, etc.).
* Subject under court protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the rate of negativation of NAATs performed at the various sites of CT infection | 4 weeks after initiation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Service du Trait d'Union, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No